CLINICAL TRIAL: NCT01017744
Title: Respiratory Mechanical Effects of Sevoflurane Administered With the Anesthetic Conserving Device in Pressure Support Ventilation
Brief Title: Pressure Support Ventilation With the Anesthetic Conserving Device
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0062
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Intensive Care Ventilation
Keywords: Anesthetic Conserving Device; Anaconda®; Sevoflurane; Remifentanil; Sedation; Pressure support ventilation; Work of breathing; Intrinsic positive end expiratory pressure; Ventilatory dead space; Intensive care; Weaning of mechanical ventilation; Ventilated ICU patients in PSV; No more in acute state; No respiratory distress; Sedated by intravenous remifentanil; In light sedation as define by a Richmond Agitation Sedation Scale (RASS) of - 1 to - 2.

INTERVENTIONS:
Device: Anesthetic Conserving Device — * Ventilation in PSV with the Anesthetic Conserving Device with remifentanil
  * Ventilation in PSV with the Anesthetic Conserving Device with sevoflurane

SUMMARY:
Sevoflurane inhalational anesthetic has got pulmonary effects such as bronchodilatation. These effects could be of interest in intensive care patients ventilated in pressure support ventilation mode. The purpose of this study is to evaluate mechanical respiratory effects of sevoflurane administered through a new specific heat and moister exchanger called the Anesthetic Conserving Device (AnaConDa®) in pressure support ventilation in intensive care patients. In fact, dead space and resistance generated by the device could cancel and even deteriorate the potential positive effects of sevoflurane on ventilation.

DETAILED DESCRIPTION:
Pharmacological sedation is often necessary in mechanical ventilated intubated patient. Since a little time, sevoflurane can be used in the intensive care unit via a specific heat and moister exchanger called the Anesthetic Conserving Device (AnaConDa®, SedanaMedical AB, Uppsala, Sweden) placed between the Y piece of the ventilatory circuit and the endotracheal tube. Sevoflurane is known to have ventilatory interesting effects such as bronchodilatation that can be useful in the treatment of severe asthma. These effects could be of interest in the intensive care ventilated patients. On the other hand, the AnaConDa® device could have negative influence on ventilatory mechanics caused by the increased dead space and the resistance to air flow. This negative effect with worsening of work of breathing (WOB) was demonstrated with classic heat and moister exchanger compared to heated humidifiers in pressure support ventilation (PSV). In this way, we would like to study the mechanical effects of the sevoflurane administered with the AnaConDa® compared to a classic management with a heated humidifier and sedation with intravenous remifentanil in PSV consecutive intensive care patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults ICU patients who are no more in acute state, intubated and ventilated in pressure support ventilation with intravenous sedation by remifentanil, with light sedation (RASS -1 to -2).

Exclusion Criteria:

* Respiratory distress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Work Of Breathing (WOB) measured during the last 5 minutes of the 20 minutes period of each treatment | during the last 5 minutes of the 20 minutes period of each treatment

SECONDARY OUTCOMES:
Intrinsic positive end expiratory pressure (PEEPi), occlusion pressure (P0,1), peak expiratory resistance, respiratory rate, tidal volume, minute ventilation, death space volume. | in PSV consecutive intensive care patients

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CONSTANTIN, General ICU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-FERRAND, Clermont-Ferrand, France

REFERENCES:
- [Background] Constantin JM, Futier E, Perbet S, Roszyk L, Lautrette A, Gillart T, Guerin R, Jabaudon M, Souweine B, Bazin JE, Sapin V. Plasma neutrophil gelatinase-associated lipocalin is an early marker of acute kidney injury in adult critically ill patients: a prospective study. J Crit Care. 2010 Mar;25(1):176.e1-6. doi: 10.1016/j.jcrc.2009.05.010. Epub 2009 Sep 24. PMID 19781900